CLINICAL TRIAL: NCT06562283
Title: Evaluation of the Reproducibility of a Fatigability Test Fitted to Patients With Spinal Muscular Atrophy
Acronym: FANTASI-SMART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 23CH295; ANSM (Other: 2024-A00225-42)
Record Dates: First submitted 2024-08-05; First posted 2024-08-20 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-11

CONDITIONS: Spinal Amyotrophy; Infantile Spinal Muscular Atrophy; Juvenile Spinal Muscular Atrophy
Keywords: Spinal Muscle Atrophy; Neuromuscular performance; Fatigue; Peripheral fatigue
MeSH Terms: conditions — Muscular Atrophy, Spinal; Spinal Muscular Atrophies of Childhood; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ambulatory patients (SMA-AMB) (Experimental): The patient is said to be "ambulant" if he or she is able to walk and perform a muscle contraction test with the quadriceps.
  Interventions: Other: Grip test; Other: Quadriceps Intermittent Fatigue test (QIF test))
- Non-ambulatory patients capable of effective grasping (SMA-PRE) (Experimental): The patient is said to be "non-ambulant", with the ability to grasp the hand.
  Interventions: Other: Thumb test; Other: Grip test
- Non-ambulatory patients without grasping ability (SMA-POU) (Experimental): The patient is said to be "non-ambulant", with the ability to contract the thumb, but without the ability to grasp the hand.
  Interventions: Other: Thumb test

INTERVENTIONS:
Other: Thumb test — Thumb adduction test consisting of intermittent, repetitive isometric contractions lasting 5 seconds at incremental percentages of maximum force.
  Arms: Non-ambulatory patients capable of effective grasping (SMA-PRE); Non-ambulatory patients without grasping ability (SMA-POU)
Other: Grip test — Muscle contraction gripping test, consisting of intermittent, repetitive isometric contractions lasting 5 seconds at incremental percentages of maximum force.
  Arms: Ambulatory patients (SMA-AMB); Non-ambulatory patients capable of effective grasping (SMA-PRE)
Other: Quadriceps Intermittent Fatigue test (QIF test)) — Quadriceps muscle contraction test consisting of intermittent, repetitive isometric contractions lasting 5 seconds at incremental percentages of maximum force.
  Arms: Ambulatory patients (SMA-AMB)

SUMMARY:
Spinal muscular atrophy (SMA) is an autosomal recessive neuromuscular disease caused by the degeneration of motor neurons in the anterior horn of the spinal cord, due to the absence of the SMN1 gene and the resulting lack of SMN protein. Some patients with particularly severe forms (types 0 or 1) die before the age of 2 in the absence of treatment, while others retain autonomous walking throughout their lives, with no reduction in life expectancy. Three treatments aimed at restoring SMN (TRS) protein expression have recently been approved by the US Food and Drug Administration and the European Medicines Agency (i.e. Nusinersen / Onasemnogene Abeparvovec / Risdiplam). Patients treated with TRS after the onset of symptoms (symptomatic patients) may show significant motor improvement, but retain difficulties such as muscle weakness and fatigue leading to limitations in activities of daily living. The aim of this study is to adapt a fatigability test, widely validated in its original version in different populations (QIF test), but adapted in this protocol to the motor level and low abilities of certain SMA patients. Our objectives are to determine whether these assessments are feasible in SMA patients, reproducible, and relevant for monitoring this population, either routinely or for future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed spinal muscular atrophy
* Age ≥ 6 years
* No orthopaedic surgery in the 6 months prior to inclusion
* Informed consent signed by the patient(s) or parent(s)/legal guardian(s) and assent of the patient
* Affiliated or beneficiary of a health insurance scheme (for inclusion in France)

Exclusion Criteria:

* Other condition that may significantly interfere with the assessment of the SMA and which is clearly unrelated to the disease
* Other associated neurological disease
* Joint deformities that prevent correct and comfortable positioning with the various different measuring devices (thumb-index clamp, handgrip and QIF-test)
* Contraindication to transcranial magnetic stimulation

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-06 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Feasibility of a fatigability test adapted to the motor level of the entire population of patients with spinal muscular atrophy. | Day : 1
  Feasibility will be assessed by the patient's success in performing the fatigability test: i.e. performing at least 2 incremental steps (i.e. at least 10 contractions at 10% of their maximum strength, then 10 contractions at 20% of their maximum strength). Validation of the feasibility of the fatigability test will be obtained if at least 80% of patients are able to perform at least the first 2 stages.

SECONDARY OUTCOMES:
Tolerance of fatigability test - Pain | Day : 1
  The tolerance of the fatigability test will be measured by a visual analogue pain scale for adults and the FPS-R face scale for children, as recommended by the French National Authority for Health (HAS)
Tolerance of fatigability test - RPE | Day : 1
  The tolerance of the fatigability test will be measured by perception of exertion (RPE) using the Borg scale (from 0 - rest to 10 - Maximal perceived effort).
Tolerance of fatigability test - AEs | Day : 1
  The tolerance of the fatigability test will be measured by the recording of adverse events (AEs) such as pain, discomfort, cramp; before, at each stage and at the end of the test.
  Tolerability of the fatigability test will be achieved if at least 90% of patients are able to carry out the test without having to stop it early because of the occurrence of AEs.
Reproducibility of the fatigability test | Day : 1
  The reproducibility of the fatigability test will be assessed by measuring and comparing the maximum voluntary force (MVC, en Nm) and the loss of force, assessed by the same assessor.
Reproducibility of the central and peripheral components of fatigue - VA | Day : 1
  The reproducibility of the central and peripheral components of fatigue will be assessed by the difference in the level of voluntary activation (% Voluntary Activation, VA) assessed by the same assessor.
Reproducibility of the central and peripheral components of fatigue - magnetic jerk | Day : 1
  The reproducibility of the central and peripheral parts of the fatigue will be evaluated by the difference in the amplitude of the magnetic jerk at rest (% jerk) of the muscles investigated, evaluated by the same evaluator.
Perceived fatigue - FACIT-F | Day : 1
  Perceived fatigue will be measured by the FACIT-F questionnaire (Functional Assessment of Chronic Illness Therapy) for adult patients. The FACIT-F is the instrument most frequently used to assess fatigue in the various chronic pathologies associated with chronic fatigue. It consists of a short questionnaire with 13 questions, which the patient answers on a scale from 0 to 4. The scores are added together, inverting the scale for negative sentences, to give a score out of 52 points. The lower the score, the greater the fatigue.
Perceived fatigue - PedsQL 4.0 | Day : 1
  Perceived fatigue will be measured by the PedsQL 4.0 fatigue questionnaire in the youngest patients (questionnaire for 6-8 year olds, 8-12 year olds, 12-17 year olds). Scores are transformed on a scale from 0 to 100, with higher scores indicating better functioning, ie lower fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard FEASSON, MD PhD, Principal Investigator — CHU SAINT-ETIENNE
Locations (4):
- France (4):
  - HCL - Hôpital Croix Rousse, Lyon
  - HFME - Hospices Civils de Lyon, Lyon
  - Aphp - Hopital Pitie Salpetriere, Paris
  - Unités de Myologie et de Médecine du Sport, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No